CLINICAL TRIAL: NCT05810597
Title: A Bioequivalence Study to Compare the Pharmacokinetics of Tirzepatide Administered Subcutaneously by a Test Device (Test Formulation) Versus Reference Device (Reference Formulation) in Healthy Participants
Brief Title: A Research Study Looking at Similarity Between Tirzepatide Versions for Different Injection Devices
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18698; I8F-MC-GPIP (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-03-31; First posted 2023-04-12 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07-01

CONDITIONS: Healthy
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Sequence 1: Tirzepatide by Single Dose Pen (SDP)/ Multi-use Prefilled Pen (MUPFP) (Experimental): Participants received a single dose of 5 milligrams (mg) tirzepatide administered subcutaneously (SC) via an SDP in Period 1 followed by a single dose of 5 mg tirzepatide administered SC via a MUPFP in Period 2.
  There was a washout period of at least 35 days between tirzepatide dose administrations.
  Interventions: Drug: Tirzepatide; Device: Single Dose Pen; Device: Multi-use Prefilled Pen
- Sequence 2: Tirzepatide by MUPFP / SDP (Experimental): Participants received a single dose of 5 mg tirzepatide administered SC via a MUPFP in Period 1 followed by a single dose of 5 mg tirzepatide administered SC via an SDP in Period 2.
  There was a washout period of at least 35 days between tirzepatide dose administrations.
  Interventions: Drug: Tirzepatide; Device: Single Dose Pen; Device: Multi-use Prefilled Pen

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
Device: Single Dose Pen — Used to administer tirzepatide SC
Device: Multi-use Prefilled Pen — Used to administer tirzepatide SC

SUMMARY:
The main purpose of this study is to look at the amount of the study drug, tirzepatide, that gets into the blood stream and how long it takes the body to get rid of it when given using two different devices. The study will also evaluate the safety and tolerability of tirzepatide and information about any side effects experienced will be collected. For each participant, the total duration of the study will be approximately 14 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant females as determined by medical history, physical examination, and other screening procedures
* Body mass index (BMI) between 18.5 and 30.0 kilograms per meter squared (kg/m²), inclusive, at screening
* Have blood pressure, pulse rate, blood and urine laboratory test results that are acceptable for the study
* Are agreeable to receiving study treatment by injections under the skin
* Are agreeable to following study contraception requirements

Exclusion Criteria:

* Have or used to have health problems that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Smoke more than the equivalent of 10 cigarettes per day
* Is a known user of drugs of abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Qps-Mra, Llc, South Miami, Florida
  - ICON Early Phase Services, San Antonio, Texas
  - ICON, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Tirzepatide by SDP / MUPFP: Participants received a single dose of 5 milligrams (mg) tirzepatide administered subcutaneously (SC) via a Single-Dose Pen (SDP) in Period 1 followed by a single dose of 5 mg tirzepatide administered SC via a Multi-use Prefilled Pen (MUPFP) in Period 2.
  There was a washout period of at least 35 days between tirzepatide dose administrations.
Period: Period 1
Arm/Group | Sequence 1: Tirzepatide by SDP / MUPFP | Sequence 2: Tirzepatide by MUPFP / SDP
Started | 34 | 31
Received At Least 1 Dose of Study Drug | 34 | 31
Completed | 31 | 31
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 1 | 0
Period: Period 2
Arm/Group | Sequence 1: Tirzepatide by SDP / MUPFP | Sequence 2: Tirzepatide by MUPFP / SDP
Started | 31 | 31
Received At Least 1 Dose of Study Drug | 31 | 31
Completed | 31 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Sequence 1: Tirzepatide by SDP / MUPFP: Participants received a single dose of 5 mg tirzepatide administered SC via an SDP in Period 1 followed by a single dose of 5 mg tirzepatide administered SC via a MUPFP in Period 2.
  There was a washout period of at least 35 days between tirzepatide dose administrations.
- Total: Total of all reporting groups
Arm/Group | Sequence 1: Tirzepatide by SDP / MUPFP | Sequence 2: Tirzepatide by MUPFP / SDP | Total
Number analyzed (Participants) | 34 | 31 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.10 (13.32) | 41.10 (14.52) | 41.10 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 16 | 14 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 33
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 29 | 29 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Tirzepatide
Description: PK: Cmax of Tirzepatide
Time Frame: Predose, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 336, and 480 hours post Day 1 dose and on Day 36 of each study period.
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Tirzepatide (SDP): Participants received 5 mg tirzepatide SC via an SDP.
- Tirzepatide (MUPFP): Participants received 5 mg tirzepatide SC via a MUPFP.
Arm/Group | Tirzepatide (SDP) | Tirzepatide (MUPFP)
Number analyzed (Participants) | 65 | 62
nanograms per milliliter (ng/mL) | 647 (31) | 524 (27)

2. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Time t, Where t is the Last Time Point With a Measurable Concentration (AUC[0-t]) of Tirzepatide
Description: PK: AUC(0-t) of Tirzepatide
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram *hour per milliliter (ng*h/mL)
Groups:
- Tirzepatide (SDP): Participants received 5mg tirzepatide SC via an SDP.
Arm/Group | Tirzepatide (SDP) | Tirzepatide (MUPFP)
Number analyzed (Participants) | 65 | 62
nanogram *hour per milliliter (ng*h/mL) | 124000 (23) | 118000 (22)

3. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of Tirzepatide
Description: PK: AUC(0-∞) of Tirzepatide
Time Frame: as for outcome 1
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tirzepatide (SDP) | Tirzepatide (MUPFP)
Number analyzed (Participants) | 65 | 61
ng*h/mL | 126000 (22) | 119000 (22)

ADVERSE EVENTS:
Time Frame: Baseline Up To 82 Days
Description: All participants who received at least one dose of study drug. Based on the planned safety analysis, adverse events were collected per the treatment received.
Arm/Group | Tirzepatide (SDP) | Tirzepatide (MUPFP)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/62
Other Adverse Events (participants affected / at risk) | 38/65 | 28/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tirzepatide (SDP) (N=65) | Tirzepatide (MUPFP) (N=62)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 10 (10) | 7 (7)
Nausea (Gastrointestinal disorders) | 16 (17) | 14 (15)
Vomiting (Gastrointestinal disorders) | 9 (9) | 7 (7)
Pain (General disorders) | 4 (4) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 17 (18) | 14 (14)
Headache (Nervous system disorders) | 10 (11) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT05810597/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT05810597/SAP_001.pdf